CLINICAL TRIAL: NCT00472316
Title: A Cluster Randomized Trial of DOTS vs DOTS Plus Active Case Finding
Brief Title: Innovative Approaches to Tuberculosis Control
Status: Completed | Type: Observational
Sponsor: Johns Hopkins University (Other)
Collaborators: Universidade Federal do Rio de Janeiro (Other)
Responsible Party: Sponsor
Other Study IDs: 2U19AI045432-06 (NIH)
Record Dates: First submitted 2007-05-10; First posted 2007-05-11 (Estimated); Last update posted 2017-08-18 (Actual); Status verified 2017-08

CONDITIONS: Tuberculosis
MeSH Terms: conditions — Tuberculosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Behavioral: Active Case Finding for Tuberculosis — Active case finding of TB in the community using community health workers

SUMMARY:
This study is designed as a cluster-randomized trial. The cluster unit is at the community level. Communities will be randomized to 1 of 2 study arms: DOTS+ACF or DOTS. Communities in the DOTS+ACF arm will receive door-to-door symptom screening of the entire population by health care workers between 2 and 4 times over a 9-month period. Those communities in the DOTS-arm will receive the current standard of care in those communities (PCF). All study communities will be receiving between 4 and 6 visits by community health workers annually as part of a program to assess and follow-up illnesses in each household. Households with ill residents will be visited more often. The intervention for this study is simply adding 3 to 5 simple questions to the current protocol. For subjects responding positively to these questions, results will be returned to the subject at their home and routine, standard of care follow-up diagnostic and treatment algorithms will be followed.

DETAILED DESCRIPTION:
Despite free ARV drugs and free TB treatment, and an expanding DOTS program, TB rates have not diminished in this city overall (29), suggesting that DOTS alone will not be sufficient to turn the tide. Nevertheless, an elemental ACF strategy did appear to work well in this city. A prior International Collaborations in Infectious Disease Research (ICIDR), in one area of Rio de Janeiro, evaluated the use of the WHO's directly observed therapy, short course (DOTS) strategy versus an enhanced DOTS strategy (DOTS-A), which included household contact investigation as a means of identifying cases. A statistically significant reduction in incidence rates between DOTS versus DOTS-A communities was seen from 2000 to 2002 (Figure 2), suggesting that ACF strategies can be instrumental in reducing incidence rates if subjects are detected and treated. Treatment completion rates among new TB cases were not significantly different statistically in the 2 study arms, however treatment completion rates overall increased from 68% to 77% over the course of the study. Overall, the DOTS communities exhibited little change (+7%) in TB incidence over the 5-year period, while DOTS-A communities showed a combined decrease (-14%) (P<0.05). The difference suggests that a large scale ACF campaign at a more intensive level (ie, door-to-door case finding) could have a significant impact on long-term TB incidence in a community.

ELIGIBILITY:
Inclusion Criteria:

* All residents of the study communities will be eligible to be surveyed at their homes, regardless of gender, age, or ethnicity.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Residents of AP3.1 and AP 5.3 in Rio de Janeiro Brazil
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Actual)
Dates: Start 2007-05; Primary Completion 2009-10 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
To compare TB incidence in communities randomized to DOTS+ACF and DOTS alone over the 18-month period following ACF campaign. | 18 months following invetervention

SECONDARY OUTCOMES:
To compare case notification rates of TB in the 2 arms of the study during the ACF campaign. | During the intervention

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Golub, PhD, Principal Investigator — Johns Hopkins University
Locations (1):
- The Health Department of Rio de Janeiro, Brazil, Rio de Janeiro, Brazil